CLINICAL TRIAL: NCT02667340
Title: Effects of Starch Produced From Heat-treated Corn (Superstarch) Supplementation on Skills, Cognitive Function and Physical Performance During/Following a Simulated Soccer Game
Brief Title: Superstarch and Physical/Cognitive Performance Following a Simulated Soccer Game
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, PhD. Weider Research Chair, University of Western Ontario, Canada
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 10009797
Record Dates: First submitted 2016-01-19; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Effect of Superstarch on Soccer Performance
Keywords: exercise; carbohydrate; Superstarch
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Superstarch (Experimental): Supplementation with Superstarch before a simulated soccer game
  Interventions: Dietary Supplement: Superstarch
- Placebo (Placebo Comparator): Supplementation with placebo before simulated soccer game.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Superstarch — 0.7 g Superstarch or placebo per kg body mass in two ingestions (before game & at halftime)
  Other Names: UCan
  Arms: Superstarch
Other: Placebo — 0.7 g glucose per kg body mass in two ingestions (before game & at halftime)
  Arms: Placebo

SUMMARY:
To assess the efficacy of a hydrothermally modified starch supplement (Superstarch made byGeneration UCAN) vs isoenergetic placebo (glucose) on exercise performance, execution of specific soccer skills, and on cognitive function during and following a simulated soccer game.

Secondary: To compare fat oxidation and carbohydrate oxidation (based on RER data) during the game with Generation UCAN vs isoenergetic placebo (glucose).

DETAILED DESCRIPTION:
This will be a double blind cross over study. There will be two treatments involved: Superstarch and glucose (placebo). Participants and investigators will be blinded as an individual not involved in the project will prepare and distribute the treatment (drinks) according to a coding system that is kept confidential until the study is completed. Participants will complete each treatment once and the treatment order will be systematically rotated to avoid any order effect. Healthy men and women soccer players aged 18-35 yr will be recruited. Participants will come to the lab on five different occasions to complete two familiarization sessions, a baseline testing session, and two main trials. During the first visit, the participants will be asked to complete a physical activity readiness questionnaire (as approved previously; Par Q and a participant information form for personal and familial health history to rule out any pathologies or health issues that may preclude them from participating in the present study. Subsequently, the investigators will collect data for VO2max, body composition and sprinting speed. In the second visit, participants will be familiarized with the high intensity intermittent exercise protocol to be used during the study days and will also be allowed to practice the cognitive and skill tests to be used (up to 8 times in order to remove any learning effect that may influence the results). During the third visit, baseline scores for the skill tests will be collected. Participants will perform 4 attempts (the first two will be for re-acclimation) and the last two will be recorded. The remaining two visits will be the study days and will be separated by at least 1 week. The order of treatments will be randomized to avoid any order effect. The night before study day, participants will arrive at the laboratory at 19:00 h and will be fed a standardized meal containing 2g/kg of carbohydrate (pasta and tomato sauce) and will not be allowed any food or drink except water thereafter. On the study day, participants will arrive to the lab at 07:30 h following an overnight 12h fast and will have refrained from exercise, caffeine or alcohol within the prior 24 hours. Baseline capillary blood lactate and blood glucose will be obtained by fingerprick by a trained phlebotomist. In order to ensure the prevention of infection and or contamination during sampling, standard sterile blood handling techniques will be used including the use of new medical examination gloves, alcohol swabs, and disposable sterile lancets. All blood-contaminated materials will be disposed of in a hazardous material labeled disposal (or sharps) container, promptly after analysis. Subsequently, baseline data for the cognitive tests will be collected. After collecting baseline data, the corresponding treatment will be given and 30 minutes after, participants will perform a standardized 10-minute warm-up, followed by the exercise session. The exercise session consists of a 60- minute simulated soccer game divided into 4 x 15-minute blocks exercising (running) at varying intensities that replicate the activity pattern of soccer such as sprinting, jogging, cruising, walking etc. The proportion of time spent at each speed will be allocated based on a time-motion analysis of professional soccer players observed by Reilly and Thomas (1976) as indicated by Clarke et al (2008). During each 15-minute block, cognitive function will be tested using the serial seven subtraction test and the Flanker test. Also, expired gas samples will be collected during the last 4 min of each standardized 15-minute block to estimate carbohydrate and fat oxidation. A fingerprick blood lactate and blood glucose sample will be collected at the end of each 15-minute block. Ratings of perceived exertion will also be taken at the end of each block. Water will be available ad-libitum during the first test day and will be quantified. The same amount of water will be provided for the remaining trial. After completion of the 60-minute simulated soccer game, we will test physical performance using a repeated sprint ability test comprised of twelve, 30m sprints with 35sec of walking recovery between each sprint. Subsequently, technical skills will be assessed using a battery test comprised of the Slalom Dribble test and the Loughborough Soccer Passing Test (LSPT). The Slalom Dribble test is a skill test that requires participants to dribble a soccer ball around a set obstacle course taking the least amount of time possible whereas the LSPT is a test that requires participants to accurately pass a soccer ball a set number of times towards coloured targets while negotiating a coned area, as quickly as possible.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female elite soccer players who are involved in regular soccer training
* aged 15-35 years

Exclusion Criteria:

* Smoker
* taking part in other research
* have a neurological or psychiatric condition that may cause cognitive dysfunction
* for women, if they are pregnant or become pregnant during the study
* Injury limiting exercise ability

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
change in exercise performance | baseline; 60 minutes later (following soccer game)
  sprint run test (seconds); soccer skills (seconds), cognitive skills (seconds)

SECONDARY OUTCOMES:
change in blood glucose concentration | baseline; 60 minutes later
  mmols/l
change in blood lactate concentration | baseline, 60 minutes later
  mmols/l

CONTACTS AND LOCATIONS:
Overall Officials: Pete W Lemon, PhD, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No